CLINICAL TRIAL: NCT06673940
Title: Effect of Transcutaneous Electrical Nerve Stimulation Applied to Acupuncture Points on Gait and Quality of Life in Stroke Patients: a Randomized Controlled Study.
Brief Title: TENS Effect on Gait and QoL in Stroke.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amina Awad,PhD, Associate Professor, Department of Physical Therapy for Neurology and Neurosurgery, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.TREC / 012 / 003990
Record Dates: First submitted 2024-10-31; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Stroke
Keywords: Stroke; spasticity; TENS; acupuncture points; gait; quality of life
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Blinded randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: stactician
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Active Comparator): TENS applied to acupuncture points in addition to physical therapy program
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS); Other: Physical Therapy program
- control arm (Active Comparator): only physical therapy program
  Interventions: Other: Physical Therapy program

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation (TENS) — TENS is applied on the acupuncture points Intervention arm
  Arms: Intervention arm
Other: Physical Therapy program — Physical therapy methods

SUMMARY:
A study was conducted to investigate the additional effect of TENS applied to acupuncture points to the physical therapy program on gait and quality of life in stroke patients.

Thirty stroke patients from both sexes aging from 40 to 65 years were randomly assigned into two equal groups: study group and control group. The study group received TENS plus the designed physiotherapy program and the control group received only the same designed physiotherapy program. The outcome measures concerned with spasticity, gait and QoL.

DETAILED DESCRIPTION:
A RCT study conducted to investigate the additional effect of TENS applied to acupuncture points to the physical therapy program on gait and quality of life in stroke patients. The study was conducted at the outpatient clinic of Faculty of Physical Therapy, Cairo University and Kasr El-Ainy Hospitals, Faculty of Medicine, Cairo University, Egypt.

Forty subjects were screened for eligibility but only thirty stroke patients from both sexes aging from 40 to 65 years who were included and randomly assigned into two equal groups: study and control group. The study group received TENS plus the designed physiotherapy program and the control group received only the same designed physiotherapy program. Patients were treated three times weekly for four weeks.

The outcome measures included the Modified Ashworth Scale (MAS) for assessing spasticity, the WHOQOL-BREF scale for evaluating QoL and the Biodex Gait Trainer for measuring the gait kinematics. Evaluation of all variables took place pretreatment and post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic stroke disease (6-8- months)
* Age 45-60 years old
* Mild to moderate spasticity
* Can walk 10 meters independently
* Sufficient cognitive abilities

Exclusion Criteria:

* Other neurological diseases
* Severe spasticity
* Cognitive impairments
* Medical instability
* Sever arthritis or contractures
* Cardio-pulmonary disorders

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth scale (MAS) | • "At baseline and at the end of treatment at 4 weeks"
  Spasticity assessment scale. Score (0-4) 0 means no increase in tone. 4 means rigidity The lower the score, the lower spasticity the patient has.
World Health Organization quality of life instrument "WHOQOL-BREF" | • ""At baseline and at the end of treatment at 4 weeks""
  Quality of life assessment questionnaire. A validated Arabic version was used. 26 items The scores on the scale from 1- 5 : 1 is the lowest score while 5 is the highest score. The higher score the participants get, the better QoL they have
Biodex Gait Trainer | • ""At baseline and at the end of treatment at 4 weeks""
  A special treadmill to measure gait kinematic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Maram A Mahmoud, MSc, Principal Investigator — Cairo University; Nahed A Salem, PhD, Study Chair — Cairo University; Ebtesam M Fahmy, PhD, Study Chair — Cairo University; Amina M Awad, PhD, Study Director — Cairo University; Asma A Salem, PhD, Study Director — Faculty of Physical Therapy Suez University; Sarah Heneidy, PhD, Study Director — Cairo University; Rania M Tawfik, PhD, Study Chair — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No